CLINICAL TRIAL: NCT01480908
Title: Postoperative Right Bundle Branch Block - Long-term Effect on the Right Ventricle in Children Operated for Ventricular Septal Defect
Brief Title: Right Bundle Branch Block After Surgical Closure of Ventricular Septal Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VSDRBBBB-RV
Record Dates: First submitted 2011-11-16; First posted 2011-11-29 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-08

CONDITIONS: Bundle-Branch Block; Heart Septal Defects, Ventricular
Keywords: Right bundle branch block; Ventricular septal defect; Echocardiography; MRI; Exercise testing
MeSH Terms: conditions — Bundle-Branch Block; Heart Septal Defects, Ventricular | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VSD, +Right bundle branch block (Experimental): Patients undergone surgical closure of ventricular septal defect and have a postoperative right bundle branch block, about 20 patients
  Interventions: Procedure: Echocardiography at rest; Procedure: Echocardiography during exercise; Procedure: MRI at rest; Procedure: Exercise testing
- VSD, -Right bundle branch block (Experimental): Patients undergone surgical closure of ventricular septal defect and does not have a postoperative right bundle branch block, about 20 patients
  Interventions: Procedure: Echocardiography at rest; Procedure: Echocardiography during exercise; Procedure: MRI at rest; Procedure: Exercise testing
- Control (Experimental): Healthy control subjects, about 20 patients
  Interventions: Procedure: Echocardiography at rest; Procedure: Echocardiography during exercise; Procedure: MRI at rest; Procedure: Exercise testing

INTERVENTIONS:
Procedure: Echocardiography at rest — Dimensions of all 4 chambers, inspiratory collapse, and gradient over the tricuspid valve is measured. Tricuspid Annulus Plane Systolic Excursion(TAPSE) and Tricuspid Annular peak Systolic Motion(TASM) is measured as well.
Procedure: Echocardiography during exercise — TASM is measured during exercise along with pulse measurements to evaluate the force-frequency-relation.
Procedure: MRI at rest — Dimensions of all 4 chambers are measured at end-systole and end-diastole. Blood flow measurements through the aortic and the pulmonary valve are made as well. No use of contrast.
Procedure: Exercise testing — Maximal oxygen consumption is measured during on a bicycle. Prior to the test a spirometry is performed to rull out potential differences in pulmonary function between the cohorts. During the test pulse, blood pressure, saturation, and EKG are monitored. Ventilatory volume, oxygen consumption and carbon dioxide excretion are measured. Anaerobic threshold is calculated at the end of the test.

SUMMARY:
The most common congenital heart disease is the ventricular septal defect, and after surgical closure of a such defect, an arrythmia called the right bundle branch block, is very frequent. Therefore the aim of this study is to investigate if this group of patients has inferior outcomes compared to the group without this arrythmia after surgical closure and compared to a group of healthy control subjects.

All patients will be undergoing 1. exercise testing, 2. echocardiography, 3. echocardiography during exercise, and 4. MRI. The perspective is the ability to point out a group of patients with a possible need of further intervention, and additionally to increase the awareness of protecting the electrical system of the heart during the operation.

DETAILED DESCRIPTION:
Right bundle branch block is an exceedingly frequent complication in heart surgery, and especially in patients who have undergone surgical closure of a ventricular septal defect which is the most common congenital heart disease. How this bundle branch block effects the right ventricle of the heart on a long-term basis for this group of patients, is still unknown.

As a part of a PhD-study we therefore will try to illustrate this by echocardiography, MRI, exercise testing and other investigations 15 to 20 years after the surgical procedure. The study population thus consists of three different groups: 1. Patients whom undergone surgical closure of ventricular septal defect without postoperative right bundle branch block, 2. VSD-operated patients with right bundle branch block and 3. Healthy controls with no significant medical issues matched on age and sex. By carrying out the tests mentioned the right ventricles systolic function, diastolic function, the patients maximal exercise capacity and a lot of other parameters will be evaluated in the three groups of patients and compared amongst each other. The perspective therefore is the ability to point out a specific group of patients with an inferior outcome and with a possible need for further intervention. An additional perspective is to increase the awareness of protecting the bundle branch during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Operated for VSD in the period from 1990 to 1995 on Aarhus University Hospital Skejby

Exclusion Criteria:

* No chart to be found
* No EKG to be found
* Known bundle branch block prior to the surgery
* Other arrythmias
* Use of ventriculotomy
* Other disease than VSD
* Pacemaker or other metallic implants
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Systolic function at rest measured by echocardiography | All patients are tested only once about 20 years post to surgery
  Dimensions of all 4 chambers, inspiratory collapse, and gradient over the tricuspidale valve is measured. Tricuspid Annulus Plane Systolic Excursion(TAPSE) and Tricuspid Annular peak Systolic Motion(TASM) is measured as well.

SECONDARY OUTCOMES:
Maximal oxygen consumption during exercise | All patients are tested only once about 20 years post to surgery
  Maximal oxygen consumption is measured during on a bicycle. Prior to the test a spirometry is performed to rull out potentiel diffenrences in pulmonary function between the cohorts. During the test pulse, blood pressure, saturation, and EKG are monitored. Ventilatory volume, oxygen consumption and carbondioxide excretion are measured. Anaerobic threshold is calculated at the end of the test.
Force-frequency-relation during exercise | All patients are tested only once about 20 years post to surgery
  TASM is measured during exercise along with pulse measurements to evaluate the force-frequency-relation.
Diastolic function at rest measured by MRI | All patients are tested only once about 20 years post to surgery
  Dimensions of all 4 chambers are measured at end-systole and end-diastole. Blood flow measurements through the aortic and the pulmonary valve are made as well. No use of contrast.
Diastolic function at rest measured by echocardiography | All patients are tested only once about 20 years post to surgery
  Dimensions of all 4 chambers, inspiratory collapse, and gradient over the tricuspidale valve is measured. Tricuspid Annulus Plane Systolic Excursion(TAPSE) and Tricuspid Annular peak Systolic Motion(TASM) is measured as well.
Systolic function at rest measured by MRI | All patients are tested only once about 20 years post to surgery
  Dimensions of all 4 chambers are measured at end-systole and end-diastole. Blood flow measurements through the aortic and the pulmonary valve are made as well. No use of contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Hjortdal, MD, DMSc, Prof., Study Chair — Dept. of Cardiothoracic surgery, Aarhus Universitetshospital Skejby; Michael R. Schmidt, MD, PhD, Study Director — Dept. of Cardiology, Aarhus University Hospital Skejby; Steffen Ringgaard, Physics, PhD, Study Director — Dept. MRI, Aarhus University Hospital Skejby; Andrew Redington, MD, DMSc, Prof., Study Director — Dept. of Cardiology, The Hospital for Sick Children, Toronto
Locations (1):
- Aarhus University Hospital Skejby, Aarhus, Aarhus N, Denmark